CLINICAL TRIAL: NCT05396456
Title: Autologous Muscle Fiber Fragment Injections for the Treatment of Fecal Incontinence
Brief Title: Autologous Muscle Fiber Fragment Injections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085606
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Fecal Incontinence
Keywords: low anal pressures; passive incontinence; bowel movements; sphincter muscle
MeSH Terms: conditions — Fecal Incontinence | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Patients with refractory Fecal Incontinence (FI) will be identified from the Atrium Wake Forest Baptist Health outpatient Gastroenterology, Urogynecology and Colorectal Surgery clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle Fiber Fragment (MFF) injections (Experimental): autologous muscle fiber fragment injections, harvested in an autologous fashion from the quadriceps muscle, for the treatment of Fecal Incontinence (FI) symptoms in men and women with a demonstrated anal sphincter defect and who have failed conservative treatments
  Interventions: Procedure: Muscle Fiber Fragment (MFF) Injections

INTERVENTIONS:
Procedure: Muscle Fiber Fragment (MFF) Injections — The participant will be treated with an injection of muscle fiber fragments into the external anal sphincter at 3, 6, 9 and 12 o'clock using a 21-gauge needle to a depth of 1-2 cm from the external skin using equal amounts in each quadrant.

SUMMARY:
To regenerate functional anal sphincter muscle using muscle fiber fragments that contain muscle precursor cells (MPCs)

DETAILED DESCRIPTION:
The Study hypothesizes that efficient re-assembly of injected fragments within host muscle tissue along the fiber direction of native muscle will be induced. It is anticipated that these fiber fragments would integrate into the host vascular and neural network.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* participants must experience 4 or more Fecal Incontinence (FI) episodes per 2 week period
* participants must score >10 on Cleveland Clinic Fecal Incontinence Severity Scoring System (CCIS)
* participants must have had symptoms for at least 12 months
* participants who have failed standard medical and surgical treatments for FI
* participant will undergo anorectal manometry (ARM) testing
* participants will undergo endoscopic anal ultrasound and demonstrate an anatomic defect of the anal sphincter complex of at least 30 degrees
* women of childbearing potential must use acceptable contraceptives during this study

Exclusion Criteria:

* participants with symptomatic anorectal disease including symptomatic hemorrhoid disease, anal fissure or fistula causing symptoms such as bleeding, swelling, pain, or drainage
* participants with pre-existing ano-rectal pain of any cause
* participants with incontinence of flatus only
* chronic watery diarrhea which is the primary cause for fecal incontinence
* acute or chronic anorectal infections (including proctitis, recurrent abscesses, fistulae)
* presence of anorectal tumors
* active proctitis or inflammatory bowel disease
* previous injection of internal anal sphincter (IAS) with bulking agents
* participants requiring immunosuppression or who have any malignant disease within 3 years of enrollment
* participants with a defined bleeding disorder diagnosed and treated by a hematologist
* other exclusions include history of pelvic radiation, rectal prolapse, anorectal malformations, anorectal surgery within the previous 12 months, or treatments using injection or infrared coagulation for treatment of hemorrhoids
* participants with neurologic disease characterized by significant peripheral neuropathy or spinal cord dysfunction
* women who are pregnant, breastfeeding, or have had a child within the last year
* participants with a history of unstable cardiac function (New York Heart Association Functional Classification III or IV) or unstable pulmonary function requiring home oxygen, or abnormal kidney function (Cr >1.5 mg/dl or on dialysis) or uncontrolled diabetes (Hemoglobin A1C > 8 mg/dl)
* participants with anemia (hemoglobin <10g, increased alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2 times normal) or increased bilirubin >1.5mg/dl
* participants with Hepatitis B or C, or human immunodeficiency virus (HIV)-1 or 2
* rectal prolapse
* vaginal prolapse beyond the hymen
* unable to understand informed consent information even with provision of a medical translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cleveland Clinic Fecal Incontinence Severity Scoring System (CCIS) scores (also termed the Wexner score) | Month 3
  fecal incontinence score from 0-20; where 0 is perfect continence and 20 is complete incontinence
Cleveland Clinic Fecal Incontinence Severity Scoring System (CCIS) scores (also termed the Wexner score) | Month 6
  fecal incontinence score from 0-20; where 0 is perfect continence and 20 is complete incontinence
Cleveland Clinic Fecal Incontinence Severity Scoring System (CCIS) scores (also termed the Wexner score) | Month 12
  fecal incontinence score from 0-20; where 0 is perfect continence and 20 is complete incontinence

SECONDARY OUTCOMES:
Change in Fecal Incontinence Quality of Life (FI-QOL) scores | baseline, Months 3 and 12
  The Fecal Incontinence Quality of Life Scale is composed of a total of 29 items; these items form four scales: Lifestyle (10 items), Coping/Behavior (9 items), Depression/Self-Perception (7 items), and Embarrassment (3 items).
Anorectal Manometry (ARM) Pressure scores | baseline, Months 3 and 12
  Low resting pressure is defined as <50 mmHg during the anorectal motility exam performed with high-resolution catheter (Given, Atlanta, GA). Normal resting pressures range from 50 to 100 mmHg.
  A flexible catheter with solid-state pressure transducers is placed in the anal canal and rectum to obtain standard pressure measurements
Internal Anal sphincter (IAS) Pressure scores | baseline, Months 3 and 12
  Typical resting pressure in a healthy volunteer is 40 to 60 mmHg
Rectal Anal Inhibitory Reflex (RAIR) Pressure scores | baseline, Months 3 and 12
  Low resting pressure is defined as <50 mmHg during the anorectal motility exam performed with high-resolution catheter (Given, Atlanta, GA). Normal resting pressures range from 50 to 100 mmHg.
  A flexible catheter with solid-state pressure transducers is placed in the anal canal and rectum to obtain Rectal Anal Inhibitory Reflex (RAIR)
Fecal Incontinence Severity Index (FISI) scores | baseline, Months 3 and 12
  Participants who score closer to 61 are likely to have their quality of life severely impacted by the fecal incontinence they suffer from.

OTHER OUTCOMES:
Anorectal endoscopic ultrasound (EUS) | Months 3 and 12
  This standard procedure is performed with a rotating rectal probe without sedation or deep sedation

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No